CLINICAL TRIAL: NCT07168382
Title: AI-Based Personalized Health and Self-Care: Investigating A Mobile Virtual Assistant to Address Health-Related Social Needs
Brief Title: AI-Based Personalized Health and Self-Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Sezgin (Other)
Responsible Party: Sponsor-Investigator, Emre Sezgin, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004369
Record Dates: First submitted 2025-08-14; First posted 2025-09-11 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Social Needs Status
Keywords: Social Needs; Chatbot; Community Resources
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chatbot Access (Experimental): These participants will receive access to the chatbot
  Interventions: Behavioral: DAPHNE Chatbot Intervention
- Standard of Care (Active Comparator): Participants will not receive access to the DAPHNE chatbot. These individuals will receive the usual HRSN screening/referral procedures at Nationwide Children's Hospital.
  Interventions: Other: Standard HRSN Screening and Referral (Usual Care)
- Health Care Providers (Experimental): All health care providers will receive access to the chatbot.
  Interventions: Behavioral: DAPHNE Chatbot Intervention

INTERVENTIONS:
Behavioral: DAPHNE Chatbot Intervention — The DAPHNE intervention consists of a conversational, AI-powered chatbot designed to identify and address health-related social needs (HRSNs) among caregivers of pediatric patients. Delivered via a secure mobile and web-based application, the chatbot facilitates natural language interactions to assess needs, generate personalized resource recommendations, and support real-time navigation to community-based services. Participants assigned to the intervention arm will have continuous access to the chatbot over a six-month period, including automated nudges, tailored prompts, and context-aware suggestions. The intervention is non-invasive and participant-driven.
  Arms: Chatbot Access; Health Care Providers
Other: Standard HRSN Screening and Referral (Usual Care) — Participants randomized to the control group will receive the standard-of-care HRSN screening and referral services as currently implemented in Nationwide Children's Hospital Primary Care Clinics. These services include in-clinic social needs assessments conducted during routine visits and referrals to internal or external resources, such as social work or care coordination teams. Participants in this group will not receive access to the DAPHNE chatbot.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to learn if the DAPHNE chatbot can improve caregiver engagement, usability, and integration of social care support tools into clinical workflows in caregivers of pediatric patients receiving care at the Nationwide Children's Hospital Primary Care Center (NCH PCC). This is a pilot randomized clinical trial.

The main questions it aims to answer are:

* Is the DAPHNE chatbot usable, acceptable, and minimally burdensome for caregivers over a 6-month period?
* Can the DAPHNE chatbot be effectively integrated into primary care provider workflows?

Researchers will compare the DAPHNE chatbot intervention arm to the standard of care control arm to see if the intervention improves caregiver-reported outcomes and provider workflow integration.

Participants that are patients will be randomly assigned to either the DAPHNE chatbot group or the standard of care group. Complete surveys assessing usability, acceptability, and burden and participate in brief qualitative interviews to share feedback on their experience.

Participants that are Primary Care providers will discuss integration of DAPHNE into clinical workflows and complete workflow integration assessments.

ELIGIBILITY:
Inclusion Criteria (Caregivers):

* Must be 18 years or older
* At least one unmet social need
* Low-income
* Currently under Medicaid/Medicare insurance or have no coverage

Inclusion Criteria (Primary Care Providers):

* Must be 18 years or older
* Must be employed at Nationwide Children's Hospital

Exclusion Criteria:

- Due to the intervention only being translated into English, non-English Speakers will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | 1 month post-baseline and 3 months post-baseline for Caregivers. Providers will complete this at baseline only.
  Survey measuring the participant usability of the chatbot on a range of 0 (lowest usability) to 100 (highest usability). Target ≥68.
Web Evaluation Questionnaire (WEQ) | 1 month and 3 months post-baseline
  Survey measuring the Caregiver's acceptability of the chatbot on a scale of 0% (lowest acceptability) to 100% (highest acceptability). Target ≥80%.
Patient Comprehension Questionnaire (PCQ) | Baseline and 3 months post-baseline
  Survey measuring the Caregiver's comprehension of the chatbot prompts and recommendations on a scale of 1 (least comprehension) to 5 (most comprehension). Target ≥ 4.
Feasibility of Intervention Measure (FIM) | Caregivers will complete at 3 months and 6 months post-baseline. Providers will complete at baseline and 6 months post-baseline.
  Survey measuring participant ratings of feasibility of the study implementation on a scale of 0% (least feasible) to 100% (most feasible). Target ≥80%.
Retention Rate | 1 month, 3 months, and 6 months post-baseline
  Percentage of participants completing follow-up assessments, measured as a percentage. Target ≥70%.
Social Determinants of Health | Caregivers will complete at baseline, 3 months post-baseline, and 6 months post-baseline.
  This questionnaire is a common instrument used in clinical settings to identify health-related social needs.

SECONDARY OUTCOMES:
User Chatbot Engagement | Continuous through 6 months post-baseline
  Measured via a log that captures total minutes participants spent using the chatbot, total number of logins, session durations, screenings completed, and number of resources accessed.
Provider Workflow Integration Expectancy | Baseline and 6 months post-baseline
  Survey measuring Provider rating of ease of chatbot workflow integration on a scale of 1 (lowest ease of integration) to 5 (highest ease of integration). Target ≥4.
Caregiver Qualitative interview | 3 months and 6 months post-baseline.
  Measured via qualitative themes. Caregivers will be interviewed about their perceptions of chatbot usability, acceptability, study procedures, and care experience.
Technical Performance Metrics | Continuously throughout 6 months of study involvement.
  Measurement of the accuracy of chatbot's responses as a percent from 0 (no accuracy) to 100 (always accurate). Target ≥70%
Perceived Research Burden Assessment (PeRBA) | 1 month, 3 months, and 6 months post-baseline.
  Survey measuring Caregiver burden related to study participation on a scale of 1 (most burden) to 5 (least burden). Target ≥4.
Recruitment rate | Continuous throughout 6 months of study involvement.
  Measurment as a percentage of total recruitment goal reached over time and dropout rate.
Caregiver Quality of Life Survey | Baseline, 3 months post-baseline, and 6 months post-baseline.
  Survey measuring caregiver-reported quality of life changes on a scale of 1 (least satisfied) to 6 (most satisfied)
Caregiver Stress Inventory | Baseline, 3 months post-baseline, 6 months post-baseline.
  Survey measuring caregiver stress levels and contributors to stress over time. Survey is a series of statements and caregivers record how much they agree with the statement on a scale of 1 (strongly disagree) to 5 (strongly agree).
Caregiver Self-Efficacy Scale | Baseline, 3 months, and 6 months post-baseline.
  Survey measuring Caregiver levels of self-efficacy in managing care and navigating resources. Survey is a series of statements and caregivers record how much they agree with the statement on a scale of 1 (strongly disagree) to 5 (strongly agree).
Resource Access Satisfaction Survey | 3 months and 6 months post-baseline.
  Survey completed by a Caregiver measuring how likely they are to recommend the intervention to someone who needs help finding health and/or social resources on a scale of 1 (least likely) to 10 (most likely).
Provider Qualitative Interview. | Baseline and 6 months post-baseline
  Health care providers will discuss their thoughts about using the app and offer opinions about the app and how it can improve.

OTHER OUTCOMES:
Provider Survey on Standard of Care | Baseline and 6 months post-baseline.
  Survey detailing providers pre-intervention standard workflows for addressing Health-Related Social Needs.
Electronic Health Record Review of Health-Related Social Needs (HRSN) Interventions | 3 months and 6 months post-baseline
  Frequency and types of HRSN interventions documented in Caregiver's EHR
Completed Health-Related Social Needs (HRSN) referrals. | 3 months and 6 months post-baseline
  Number of HRSN referrals completed by Caregiver (e.g., social services, specialty care).
Primary Care Visit Completion. | 3 months and 6 months post-baseline
  Percentage of completed primary care visits (i.e., Caregiver visit adherence).
Missed Appointments | 3 months and 6 months post-baseline.
  Number of caregiver missed/no-show clinic visits
Emergency Department Visits | 3 months and 6 months post-baseline
  Number of Emergency Department Visits per Caregiver
Healthcare Cost Avoidance | 3 months and 6 months post-baseline
  Estimated cost avoidance from improved visit adherence and reduced ED utilization. Reported by Caregivers in USD.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Sezgin, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Sezgin E, Clarkson E, Logan F, Jackson DI, Hussain SA, Stokes J, Bunger A, Brock G, Fosler-Lussier E, Kemper AR, Pai AL. An AI-Based Chatbot to Support Health-Related Social Needs among Pediatric Primary Care Population: Protocol for a Pilot Randomized Controlled Trial. medRxiv [Preprint]. 2025 Nov 19:2025.11.17.25340433. doi: 10.1101/2025.11.17.25340433. PMID 41332826